CLINICAL TRIAL: NCT01411904
Title: A Novel Magnetic Needle Using Iron Oxide Nanoparticles for the Detection of Leukemia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The NPs that we have been buying from a vendor show lot to lot variation. We are making our own NPs, need to characterize them before we enroll new patients.
Sponsor: University of New Mexico (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Richard Larson, Executive Vice Chancellor Vice Chancellor for Research, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-049; 5R44CA105742-05 (NIH)
Record Dates: First submitted 2011-04-18; First posted 2011-08-08 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Leukemia
Keywords: Leukemia; magnetic needle; magnetic nanoparticles; CD34
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MagProbe (TM) (Experimental): Patients whose bone marrow aspirates are exposed to the MagProbe and CD34 nanoparticles.
  Leukemia patients
  * MagProbe (TM)
  * Diagnosed or suspected leukemia
  Non-leukemia patients
  * MagProbe (TM)
  * Requiring bone marrow biopsy
  Interventions: Device: MagProbe (TM)

INTERVENTIONS:
Device: MagProbe (TM) — CD34 nanoparticles incubated in bone marrow and then extracted with the magnetic needle done at time of bone marrow biopsy
  Other Names: Magnetic Needle

SUMMARY:
The purpose of this study is to determine if the magnetic needle, in combination with magnetic nanoparticles can accurately identify minimal residual disease in leukemia patients.

DETAILED DESCRIPTION:
The ability to reliably detect Minimal Residual Disease (MRD) in leukemia patients allows oncologists to predict patient outcome and to monitor the efficacy of therapy which is critical to improving care. MRD can be used to identify high risk patients who cannot be identified by conventional high risk features, a presence of < 0.1% MRD has been shown to be one of the best predictors of 5-year remission, with 70% of patients with ≥ 0.1% relapsing. In addition to providing predictions of relapse, MRD has been shown to provide a sensitive measure of early treatment response, an independent predictor of good outcome. While the presence of MRD is indicative of patient outcome, the detection of the presence of MRD provides an opportunity to modify treatment and potentially increase survival. Studies are currently underway to use MRD detection in modifying chemotherapeutic treatment and timing of stem cell transplant in leukemia patients. Development of a low cost and easily accessible MRD detector has the potential to expand the number of patients for which MRD testing is available. Expansion of the patient population is a necessary step to large scale testing of MRD detection as both a predictive factor of patient outcome and as a potential modifier of patient treatment. It is expected that increased MRD testing would lead to improved prediction of patient outcomes and increased sensitivity of testing of treatment response. MRD testing in the general patient population could be used to test treatment response and allow oncologists to modify treatment regiments leading to reduced patient mortality and improved medical outcomes.

ELIGIBILITY:
Group: Leukemia Patients

Inclusion Criteria:

* Suspected diagnosis of Leukemia
* Requiring bone marrow biopsy for standard care

Exclusion Criteria:

* unable to consent for entrance into the study

Group: Non-leukemia Patients

Inclusion Criteria:

* Requiring bone marrow biopsy for standard care

Exclusion Criteria:

* unable to consent for entrance into the study
* Leukemia diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Lymphoblast percent | 1 day
  Lymphoblast percent calculated before exposure to needle and of the needle enhanced sample

SECONDARY OUTCOMES:
SQUID magnetometry | 1 day
  Magnetic Signal from the nanoparticles bound to the leukemia cells

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States